CLINICAL TRIAL: NCT03118752
Title: Pragmatic Collaborative Care for Cardiac Inpatients With Depression or Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Jeff C. Huffman, MD, Associate Chief of Psychiatry, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016P002870; 1R01HL133149-01A1 (NIH)
Record Dates: First submitted 2017-04-06; First posted 2017-04-18 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Acute Coronary Syndrome; Heart Failure; Depression; Generalized Anxiety Disorder; Panic Disorder
MeSH Terms: conditions — Acute Coronary Syndrome; Heart Failure; Depression; Generalized Anxiety Disorder; Panic Disorder

STUDY DESIGN:
Intervention Model Description: This study will be a randomized, controlled, 2-arm, single blinded trial.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Collaborative Care (Experimental): Participants randomized to collaborative care (CC) will receive a 26-week, telephone based CC intervention. Care managers will monitor participants' psychiatric symptoms, review current treatments for their psychiatric and cardiac illnesses, deliver psychotherapeutic interventions, provide education about self-monitoring for cardiac symptoms, perform motivational interviewing to encourage health behavior adherence, and coordinate care between psychiatric/cardiac specialists and participants' primary care physicians. CC will utilize a treat-to-target approach, with a goal of remission of psychiatric and cardiac symptoms.
  Interventions: Behavioral: Collaborative Care
- Enhanced Usual Care (No Intervention): Participants in the enhanced usual care (eUC) arm will not receive any specific intervention, though they will be free to receive any treatment for psychiatric or cardiac illness. Participants' outpatient providers will be informed of their psychiatric diagnosis, which may lead to higher-than-usual treatment for psychiatric illness.

INTERVENTIONS:
Behavioral: Collaborative Care — The CC intervention will use a novel three-pronged approach to these high-risk patients. Care managers will provide centralized care coordination and specific interventions targeting: (1) the psychiatric disorders, (2) cardiac health behaviors, and (3) the cardiac illness.
  Arms: Collaborative Care

SUMMARY:
The investigators will complete a pragmatic randomized trial (N=260 randomized participants) of the 26-week blended collaborative care (CC) intervention compared to enhanced usual care (eUC) in patients admitted for acute coronary syndrome (ACS) or heart failure (HF) found to have current depression, generalized anxiety disorder (GAD), or panic disorder (PD). The CC intervention will use a novel three-pronged approach to these high-risk patients. Care managers will provide centralized care coordination and specific interventions targeting: (1) the psychiatric disorders, (2) cardiac health behaviors, and (3) the cardiac illness. The primary study outcome will be physical function at 26 weeks, measured by the Duke Activity Status Index (DASI), given links between function and new cardiac events. The investigators will also examine effects on numerous other outcomes important to patients and healthcare systems.

Specific Aim 1 [patient-centered outcomes-primary aim]: To compare between-group differences in the CC and eUC conditions on improvements in physical function, health-related quality of life, mental health, patient satisfaction, and other key patient-reported outcomes at 26 and 52 weeks.

Specific Aim 2 [adherence and medical outcomes]: To compare between-group differences on health behaviors (physical activity, diet, smoking, medication adherence) and major adverse cardiac events.

Specific Aim 3 [cost]: To compare healthcare costs between groups and assess the cost-effectiveness of CC.

Hypotheses: The investigators expect this bolstered CC program to be associated with superior improvements in physical function, health-related quality of life, patient satisfaction, and adherence at 26 weeks, with promising effects on major adverse cardiac events. The investigators likewise expect the intervention to be cost-effective (<$10,000/quality-adjusted life year) over the study period.

DETAILED DESCRIPTION:
Study Visits/Contacts/Interventions

Procedures for Participants in the Collaborative Care Intervention

In the hospital, participants randomized to CC will work with the care manager to: (a) define specific goals related to their psychiatric condition, health behaviors, and self-care, (b) initiate care for their psychiatric condition, and (c) make a plan for a health goal, using a structured tool based on prior work, with a specific and systematic focus on social, functional, financial, and other barriers to behavior change.

Following discharge, all contact will be via phone, with the same care manager completing phone sessions to enhance alliance and care continuity. Contacts will last typically 30-45 minutes using a structured but highly flexible approach designed to manage acute issues and cover some aspect of all three care targets based on patient needs/preferences, without requiring care managers to complete all possible interventions at each call. Care managers will prioritize topics to be addressed at each contact, responding first to urgent concerns (e.g., chest pain, suicidal ideation). Next, the care manager will touch on all three aspects of the intervention, with the depth of focus for each component based on prior sessions and current issues. He/she will review psychiatric symptoms and treatment. The care manager will gauge progress on health behavior goals, review motivation/barriers to goal completion, and make an action plan for the next week. Finally, he/she will compare cardiac medication lists to guidelines and review weight/blood pressure self-monitoring. Calls will occur weekly for the first 6 weeks, then may be spaced out in subsequent weeks based on the patient's psychiatric symptoms, progress toward health behavior goals, and cardiovascular status. Both the participant and care manager will agree upon the amount of time between calls after the first 6 weeks, though participants will be encouraged to contact the care manager sooner if needed.

* 1 Targeting multiple psychiatric conditions. First, the care manager will assist in the assessment and management of depression, GAD, and/or PD using standardized scales. At weekly team meetings, care managers and supervising clinicians will review participants' scores to allow iterative recommendations for treatment, and supervision will be provided to care managers about psychotherapeutic content. A treat-to-target approach will be used for psychiatric disorders, with a goal of remission. Treatments for mood/anxiety disorders may include medications (with selective serotonin reuptake inhibitors [SSRIs] typically recommended), psychotherapy (telephone-delivered cognitive behavioral therapy [CBT] sessions, supplemented by CBT workbooks), or relaxation response (RR) training.
* 2 Targeting cardiac health behaviors. The investigators will systematically target health behaviors, primarily via motivational interviewing given its efficacy for a wide variety of behaviors in medical patients. The investigators will focus on four specific health behaviors (diet, exercise, smoking, and medication adherence). During admission, care managers and participants will identify one behavior to target and set a specific goal aligned with ACS/HF guidelines and the medical team's recommendations. Care managers will utilize motivational interviewing techniques to assist participants in considering, making, and maintaining change toward that goal. A focus on health behaviors will then continue throughout the 26 weeks.
* 3 Targeting the cardiac condition. First, care managers will review the participant's medication regimen and compare it to published guidelines for ACS and HF. The care manager will discuss this with the study cardiologist and, if the regimen appears suboptimal, they will suggest to the patient's physician(s) possible adjustments. Second, care managers will encourage participants to check blood pressure and weight daily and will review data at study calls; if the readings deviate from targets (e.g., HF patient gaining weight), the care manager will review with the cardiologist and contact patients' medical providers as indicated. The investigators will provide (commercially-available) digital scales or automated blood pressure cuffs to participants (in either group) who need them.

Procedures for Participants in Enhanced Usual Care.

For participants randomized to eUC, baseline psychiatric and medical assessments will be transmitted to the patient's electronic health record. During the enrollment admission, the care manager will also inform the participant and treatment team about the specific symptoms on the study instruments and their clinical relevance (and will alert teams to the data transmitted to the electronic health record). eUC participants also will be free to receive any treatment for mental health or cardiac conditions throughout the study.

At follow-up study assessments for eUC (and CC) participants at 26 and 52 weeks, psychiatric symptom data will be transmitted to the electronic health record, and providers will be alerted if psychiatric symptoms persist. If acute safety concerns are identified at follow-ups or other contacts, the study team will also arrange as-needed urgent care). Finally, the investigators will provide eUC participants with blood pressure cuffs and/or scales if needed, to ensure that outcome improvements in CC are not simply due to their provision.

Study Endpoints.

Functional, HRQoL, psychological, and care process outcomes (Specific Aim 1) The investigators will assess the intervention's impact on multiple functional and psychological outcomes, including physical function (using the Duke Activity Status Index (primary study outcome), generic HRQoL (Medical Outcomes Study SF-12), disease-specific HRQoL (Kansas City Cardiomyopathy Questionnaire, Seattle Angina Questionnaire), depression (SCL-20), anxiety (Hospital Anxiety and Depression Scale - anxiety subscale), optimism (Life Orientation Test - Revised), and participant satisfaction.

Behavioral and medical outcomes (Specific Aim 2) The investigators will assess the intervention's impact on adherence to medications (using the self-report medication adherence tool from the NHLBI Heart and Soul study), diet (using the MEDFICTS (meats, eggs, dairy, fried foods, fat in baked goods, convenience foods, fats added at the table, and snacks) scale for saturated fat intake and the Scored Sodium Questionnaire for sodium intake), physical activity (using the International Physical Activity Questionnaire), and smoking (7-day point prevalence smoking assessment). The investigators also will monitor for major adverse cardiac events (defined as admission for an ACS, percutaneous intervention, or acute HF, or mortality).

Cost and related outcomes (Specific Aim 3) Finally, the investigators will monitor medical utilization using Partners Healthcare records ahd the Massachusetts All Payer Claims Database. For cost effectiveness, the investigators will use the EuroQol five dimensions questionnaire (EQ-5D) health utilities scale, which allows direct assessment of cost per quality-adjusted life year.

ELIGIBILITY:
Inclusion Criteria:

1. Adults with a primary medical provider in the Partners Healthcare System admitted to Massachusetts General Hospital (MGH) or Brigham and Women's Hospital (BWH).
2. Admission for acute coronary syndrome (myocardial infarction or unstable angina) or acute heart failure.
3. Clinical depression, GAD, or PD, identified using the Patient Health Questionnaire-9 (PHQ-9) for depression and the Primary Care Evaluation of Mental Disorders (PRIME-MD) anxiety modules.

Exclusion Criteria:

1. Medical conditions precluding interviews or likely to lead to death within 6 months (per clinical team).
2. Inability to participate in study procedures: cognitive deficits (via 6-item cognitive screen designed for research) or non-fluency in English.
3. Complex psychiatric conditions. The investigators will exclude patients with bipolar disorder, psychosis, or an active substance use disorder, as well as those with active suicidal ideation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2024-03-08 (Actual); Study Completion 2024-03-08 (Actual)

PRIMARY OUTCOMES:
Change in physical function | Baseline, 26 weeks, 52 weeks
  Physical function will be assessed with the Duke Activity Status Index (DASI).

SECONDARY OUTCOMES:
Change in generic health-related quality of life | Baseline, 26 weeks, 52 weeks
  Generic HRQoL will be assessed via the Medical Outcomes Study SF-12 (SF-12).
Change in disease-specific health-related quality of life | Baseline, 26 weeks, 52 weeks
  Disease-specific HRQoL, measured via the Kansas City Cardiomyopathy Questionnaire (KCCQ; for participants with heart failure) or the Seattle Angina Questionnaire (SAQ; for participants who experienced an acute coronary syndrome).
Change in mental health (depression) | Baseline, 26 weeks, 52 weeks
  Depression will be measured by the 20-item Symptom Checklist Depression Scale (SCL-20).
Change in mental health (anxiety) | Baseline, 26 weeks, 52 weeks
  Anxiety will be measured by the Hospital Anxiety and Depression Scale, Anxiety Subscale (HADS-A).
Change in optimism | Baseline, 26 weeks, 52 weeks
  Optimism will be assessed via the well-validated Life Orientation Test-Revised (LOT-R)
Change in patient satisfaction | Baseline, 26 weeks, 52 weeks
  Participant satisfaction with mental health care and cardiac care will both be measured using 10-point Likert scales.
Change in physical activity adherence | Baseline, 26 weeks, 52 weeks
  Physical activity adherence will be measured by a 7-day physical activity recall assessment for physical activity using the International Physical Activity Questionnaire (IPAQ).
Change in dietary adherence (saturated fat) | Baseline, 26 weeks, 52 weeks
  Dietary adherence will be measured by assessing saturated fat using the MEDFICTS scale calibrated to American Heart Association guidelines.
Change in dietary adherence (sodium intake) | Baseline, 26 weeks, 52 weeks
  Dietary adherence will be assessed by sodium intake measured using the Scored Sodium Questionnaire (SSQ).
Change in smoking | Baseline, 26 weeks, 52 weeks
  Change in smoking will be measured by a 7-day point prevalence smoking assessment.
Change in cardiac medication adherence | Baseline, 26 weeks, 52 weeks
  Cardiac medication adherence will be assessed using the self-report medication adherence tool from the NHLBI Heart and Soul study.
Major adverse cardiac events | 52 weeks
  Major adverse cardiac events (MACE) will be defined as admission for an acute coronary event (ACS or new percutaneous intervention) or acute HF, or mortality.
Healthcare costs | 52 weeks
  Direct program costs will be measured by a compiled value from the following parts: (1) patient assessment (including Electronic Health Record [EHR] alerts/PROM); (2) care manager and other team member time (including training); (3) medications for psychiatric and cardiac conditions; (4) care registry development/maintenance; and (5) mental health specialty referrals. Patient costs include both direct costs (e.g., copayments) and indirect costs (patient time, valued via Bureau of Labor Statistics).
Cost-effectiveness | 52 weeks
  Cost effectiveness will be measured using the EQ-5D health utilities scale, which allows direct assessment of cost per quality-adjusted life year (QALY).

CONTACTS AND LOCATIONS:
Overall Officials: Jeff C Huffman, MD, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Salem Hospital, Salem, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The investigators will download final research data, from which the investigators will generate deidentified datasets that are free of patient names, medical record numbers, addresses, or other personal identifiers. The investigators will also review the data to ensure that there is not additional information by which patients could be deductively identified. Data will be provided in a Microsoft Excel spreadsheet or in a file compatible with specific commonly used statistical packages (Stata, SPSS, and SAS). It will be deposited in the publicly available Dataverse repository used within the Harvard system.